CLINICAL TRIAL: NCT00626353
Title: Interdisciplinary Home Rehabilitation of Patients With Stroke. A Randomised Controlled Intervention Trial.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Gentofte, Copenhagen (Other)
Collaborators: Ministry of the Interior and Health, Denmark (Other Government)
Responsible Party: Principal Investigator, Rune Skovgaard Rasmussen, PhD, MA, PhD, University Hospital, Gentofte, Copenhagen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: H-A-2007-0027
Record Dates: First submitted 2008-02-20; First posted 2008-02-29 (Estimated); Last update posted 2014-03-18 (Estimated); Status verified 2014-03

CONDITIONS: Acute Stroke
Keywords: Stroke; rehabilitation; motor recovery; cognition; quality of life
MeSH Terms: conditions — Stroke | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention (Experimental): Patients treated by an interdisciplinary, intersectoral and interventional team responsible for providing home-based rehabilitation.
  Interventions: Other: Home-based rehabilitation
- Control (Active Comparator): Control patients treated following standard care procedures in our department with no interference from the interventional team.
  Interventions: Other: Standard care

INTERVENTIONS:
Other: Home-based rehabilitation — Rehabilitation at home during hospital stay and after discharge
  Other Names: Rehabilitation at home
  Arms: Intervention
Other: Standard care — Standard care during hospital stay and in the municipality after discharge
  Other Names: Regular rehabilitation stroke treatment
  Arms: Control

SUMMARY:
Objective: To evaluate the effect of interdisciplinary home rehabilitation of patients with acute stroke. The trial seeks to evaluate:

1. Can early home rehabilitation affect the degree of independence (motor capacity, activities of daily living and cognitive status), quality of life and the possibility of discharge to own home?
2. Can home rehabilitation influence the length of admission at a rehabilitation centre in the municipality, readmission to hospital, the use of healthcare services and death?
3. To what extend can home rehabilitation be implemented according to finances? Materials and methods: Patients at the age 18 years or more admitted to the stroke unit at the University Hospital of Gentofte. The patients were eligible when meeting the following criteria: symptoms of stroke, need of rehabilitation tree days after admission, living in own home in the Municipality of Gentofte, Lyngby-Taarbaek or Rudersdal and Modified Rankin Score between 0 and 3.

The trial was conducted as a randomised controlled trial. The control group patients were rehabilitated according to normal procedure. The intervention group patients were rehabilitated according to normal procedure and were additionally rehabilitated at home during admission and four weeks after discharge.

DETAILED DESCRIPTION:
Objectives were to assess the efficacy of home-based stroke rehabilitation compared to standard care in stroke patients using an interventional, randomised, safety/efficacy open-label trial and parallel assignment. The setting was single-center, stroke unit at the University Hospital of Copenhagen, Gentofte, although patients were recruited through a collaboration of several municipalities.

Participants were eligible patients with a clinical diagnosis of stroke and focal neurological deficits hospitalised in a stroke unit for more than three days and in need of rehabilitation.

Interventions patients were randomised to home-based rehabilitation during hospitalization and for up to 4 weeks after discharge to replace part of usual treatment and rehabilitation services. Control patients received treatment and rehabilitation following usual guidelines for the treatment of stroke patients.

Main outcome measures 90 days post-stroke, modified Rankin Scale, and motor rehabilitation, cognitive abilities, quality of life and treatment-associated economy as secondary outcomes.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or more,
* Symptoms of stroke,
* Need of rehabilitation tree days after admission,
* Living in own home,
* Modified Rankin Score between 0 and 3

Exclusion Criteria:

* Terminal care,
* Discharged from another department, Living in nursery home,
* Can not understand the Danish language,
* Memory difficulties

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2007-07; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
modified Rankin Scale | 90 days
  To investigate differences in the modified Rankin Scale among intervention and control patients at the inclusion time point and 90 days later.

SECONDARY OUTCOMES:
EuroQol-5D™ quality of life measurement | 90
  To measure differences of perceived quality of life in the EuroQol-5D™ quality of life test (EQ-5D) among intervention and control patients at the inclusion time point and 90 days later.
Barthel-100 Index | 90
  To investigate differences in the Barthel-100 Index scores among intervention and control patients at the inclusion time point and 90 days later.
Motor Assessment Scale | 90
  To investigate differences in Motor Assessment Scale test scores among intervention and control patients at inclusion time point and after 90 days.
CT-50 Cognitive Test | 90
  To investigate differences in CT-50 Cognitive Test scores among intervention and control patients at inclusion time point and after 90 days.

OTHER OUTCOMES:
Body Mass Index | 90
  To investigate differences in Body Mass Index (BMI) scores among intervention and control patients at inclusion time point and after 90 days.
Economy | 90
  To estimate differences in treatment associated costs among intervention and control patients at inclusion time point and after 90 days.

CONTACTS AND LOCATIONS:
Overall Officials: Finn Roenholt, PhD, Study Director — University Hospital of Copenhagen, Gentofte Hospital
Locations (1):
- University hospital of Gentofte, Hellerup, Denmark